CLINICAL TRIAL: NCT02838745
Title: Phase I Study of Cytoreductive Surgery and Hyperthermic Intraoperative Chemotherapy With Pemetrexed and Cisplatin for Malignant Pleural Mesotheliomas
Brief Title: Study of Cytoreductive Surgery and Hyperthermic Intraoperative Chemotherapy With Pemetrexed and Cisplatin for MPM
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Change in research plan.
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Shawn Groth, Assistant Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H-36460
Record Dates: First submitted 2016-07-16; First posted 2016-07-20 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Mesothelioma
MeSH Terms: conditions — Mesothelioma | interventions — Pemetrexed; Cisplatin

ARMS (2):
- Pemetrexed (300 mg/m2) and Cisplatin (175 mg/m2) (Experimental): Pemetrexed and cisplatin will be admixed together in 1 liter of normal saline. The admixture of pemetrexed/cisplatin is stable for 4 hours and should be prepared and delivered immediately before use in the OR. The length of the pemetrexed/cisplatin lavage will be 1 hour.
  Interventions: Drug: Pemetrexed; Drug: Cisplatin
- Pemetrexed (400 mg/m2) and Cisplatin (175 mg/m2) (Experimental): Pemetrexed and cisplatin will be admixed together in 1 liter of normal saline. The admixture of pemetrexed/cisplatin is stable for 4 hours and should be prepared and delivered immediately before use in the OR. The length of the pemetrexed/cisplatin lavage will be 1 hour.
  Interventions: Drug: Pemetrexed; Drug: Cisplatin

INTERVENTIONS:
Drug: Pemetrexed
Drug: Cisplatin

SUMMARY:
Primary Objective

To determine the maximum tolerated dose (MTD) of intrathoracic administration of pemetrexed when given in conjunction with cisplatin in patients with resectable malignant pleural mesothelioma MPM.

Secondary Objectives

To determine the toxicity and grades associated with cytoreductive surgery and Hyperthermic Intraoperative Chemotherapy HIOC with cisplatin and pemetrexed in patients with resectable MPM.

To assess overall survival and progression-free survival after PD or EPP and HIOC with cisplatin and pemetrexed for MPM

Correlative Objectives

To characterize the pharmacokinetics and pharmacodynamics of pemetrexed when administered as a hyperthermic intrathoracic lavage after PD or EPP

To determine whether the degree of thymidylate synthase and ERCC1 gene expression in MPM tissue correlates with clinical response to pemetrexed.

DETAILED DESCRIPTION:
TREATMENT PLAN

PREOPERATIVE HYDRATION According to our observations, preoperative hydration reduces the risk of nephrotoxicity from intrathoracic infusion of hyperthermic cisplatin. Therefore, all patients will be admitted the night before surgery and receive intravenous hydration.

CYTOREDUCTIVE SURGERY

Eligible patients will undergo an extrapleural pneumonectomy (EPP) or pleurectomy/decortication (PD) by a Baylor College of Medicine board-certified thoracic surgeon. Patients will be given ondansetron 8mg x 1 dose after induction of anesthesia, before initiation of chemotherapy lavage. The anti-emetics will be adjusted if grade III toxicity is still encountered. Patients will then undergo cytoreductive surgery (PD or EPP) with curative intent. In the event that not all of the tumor can be removed then the investigators will allow a total of 1 cm3 or less of disease in one or more areas. If the tumor is unresectable and debulking cannot be obtained, then the patient will receive additional treatment off protocol. Mediastinal lymph node sampling will be performed. In the event that the diaphragm and pericardium are resected, they will be reconstructed with polytetrafluoroethylene (PTFE).

RENAL PROTECTION STRATEGY

The investigators will continue our established perioperative renal protection strategy to minimize the risk of cisplatin-induced nephrotoxicity.

Perioperative Intravenous Hydration:

The patient will be admitted the night before surgery for intravenous hydration.

During the operation, the anesthesiologist will monitor urine output. At his or her discretion, diuretics, renal dose dopamine, or fluid challenge will be instituted to maintain the urine output at least 100 cc per hour.

In the immediate postoperative setting, the patient will be aggressively hydrated; a pulmonary artery catheter will be used to guide management. Cisplatin-induced diuresis (more than 100 cc per hour) will be replaced with crystalloid for the first 24 hours after surgery at the following rate: 1cc crystalloid per 1cc of urine after PD and 0.5cc crystalloid per 1cc of urine after EPP.

Amifostine and Sodium Thiosulfate Per Protocol.

HEATED INTRAOPERATIVE CHEMOTHERAPY PERFUSION

The procedure is as follows:

* After the cancer resection is complete, the perfusion cannulae will be placed within the open hemithorax.
* A total of three temperature probes will be placed within the hemithorax or upper abdomen (via the chest since the diaphragm is no longer present after most PDs and after all EPPs) and the esophagus.
* Another two temperature probes will be used to monitor the temperature of the solution in the circuit.
* An open well will be created over the thoracotomy using an Omni tract retractor, using monofilament suture between the skin edges and the retractor, and enclosing the area with a plastic covering.
* A slit in the plastic cover is made just large enough to allow the surgeon's double-gloved hand into the hemithorax to evenly distribute the perfusate. The surgeon gently (but repeatedly) manipulates all exposed areas to allow uniform distribution of the heated chemotherapy.
* Pemetrexed and cisplatin will be admixed together in 1 liter of normal saline. The admixture of pemetrexed/cisplatin is stable for 4 hours and should be prepared and delivered immediately before use in the OR. The length of the pemetrexed/cisplatin lavage will be 1 hour.
* A roller pump forces the heated chemotherapy into the chest and abdomen through the inflow cannula and pulls it out via an outflow cannula.
* If the perfusate solution does not fill the chest cavity, one or more intact bags of saline will be placed in the chest cavity to displace the perfusate. In this manner, the chest cavity can be filled without diluting the perfusate.
* A heat exchanger keeps the fluid being infused at 43-45 degrees Celsius so that the intrathoracic fluid is 42 degrees Celsius.
* A smoke evacuator is used to pull air from beneath the plastic cover through activated charcoal, preventing any possible contamination of air in the operating room by chemotherapy aerosols.

Pharmacokinetics will be drawn per protocol.

Dose Levels

Cohort Pemetrexed Dose A 300 mg/m2 B 400 mg/m2 C 500 mg/m2 D 600 mg/m2 E 700 mg/m2 F 800 mg/m2 Stop to Analyze Safety G 900 mg/m2 H 1000 mg/m2 Stop to Analyze Safety

The standard dose of pemetrexed for systemic administration is 500 mg/m2. However, because pemetrexed has not been previously studied for direct administration into the chest, the initial cohorts will receive a slightly lower dose to ensure this method of administering pemetrexed is safe. Once safety has been established at lower doses, the investigators will feel confident that pemetrexed intrathoracic doses that are slightly higher than the standard systemic dose (500 mg/m2) can be given safely. In animal models, these higher doses resulted in a systemic concentration of pemetrexed (which is correlated with systemic toxicities) that is potentially lower after intracavitary infusion than after systemic administration 2. These higher doses may result in superior long-term clinical outcomes.

Schedule Assignment for Dose Levels

Patients will be enrolled in cohorts of 3 according the dose escalation/de-escalation rules specified. For the purposes of executing the dose escalation scheme, toxicity will be assessed until 4 weeks after treatment. Additional patient cohorts will not be enrolled until all toxicity evaluable patients treated at the current dose have completed the observation period. In addition, the investigators will pause after completion of the 800 mg/m2, if the MTD is not reached, to assure that delayed toxicities don't manifest. If the MTD is not exceeded at the highest dose level, the escalation schedule may be expanded.

Dose limiting toxicity (DLT) is defined as:

* Grade 4 treatment-related hematologic toxicity that lasts more than for 5 days or grade 3 thrombocytopenia with grade 3 or 4 bleeding
* Febrile neutropenia
* Grade 3 or greater treatment related non-hematologic toxicity with the following exceptions:

  * Grade 3 diarrhea is a DLT only if the patient was compliant with an anti-diarrheal program consistent with best clinical practice
  * Grade 3 or 4 nausea and vomiting is a DLT only if the patient was compliant with an antiemetic program consistent with best clinical practice
  * Alopecia

Supportive Care Guidelines All supportive measures consistent with optimal patient care will be given throughout the study.

Duration of Therapy

Patients will receive protocol therapy unless:

1. Extraordinary medical circumstances: If at any time the constraints of this protocol are detrimental to the patient's health, protocol treatment will be discontinued
2. Patient withdraws consent
3. There is evidence of progressive disease or unacceptable toxicity
4. The treating physician thinks a change of therapy would be in the best interest of the patient

Follow-up All patients, including those who discontinue protocol therapy early, will be followed by their oncologist or primary care providers. The date of death will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven malignant pleural mesothelioma MPM that is considered resectable according to the following criteria:

   * Confined to one pleural space
   * No chest wall invasion
   * No transdiaphragmatic involvement
   * No invasion of mediastinal structures
2. Age ≥ 18 years
3. Eastern Cooperative Oncology Group performance status 0-1 (Appendix A)
4. Adequate cardiopulmonary reserve defined as follows as assessed within 4 months of study entry:

   * Predicted postoperative forced expiratory volume FEV1 > 1L
   * Normal left ventricular function (Ejection Fraction EF ≥ 45%) and right ventricular function
   * No pulmonary hypertension noted on preoperative transthoracic echocardiography
5. Must have adequate hematologic, renal and hepatic function as defined by the following laboratory values (completed within 60 days of surgery) Hematologic: Hemoglobin ≥ 9.0 g/dL, absolute neutrophil count (ANC) ≥ 1500/mm3, platelet count ≥ 100,000/mm Renal: Calculated creatinine clearance ≥ 60 mL/min

   The creatinine clearance CrCl is determined by the Cockcroft-Gault formula:

   Males:

   Creatinine Clearance CrCl (mL)/min) = weight (kg) x (140-age) 72 x serum creatinine (mg/dL)

   Females:

   Creatinine Clearance CrCl (mL)/min) = weight (kg) x (140-age) x 0.85 72 x serum creatinine (mg/dL)

   Hepatic: Total bilirubin < 1.5 times the upper limit of institutional normal value; Aspartate aminotransferase AST (Serum glutamic oxaloacetic transaminase SGOT) and alanine aminotransferase ALT (Serum glutamic pyruvic transaminase SGPT) < 3 times the upper limit of the institutional normal Coagulation: international normalized ratio INR ≤ 1.5 in patients not utilizing systemic anticoagulation as part of their medical regimen
6. Women of child bearing potential and sexually active males must use an accepted and effective non-hormonal method of contraception
7. Patients must be deemed by the investigators to be fully recovered from both acute and late effects of any prior surgery, radiotherapy, or other antineoplastic therapy
8. Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
9. The ability to interrupt non-steroidal anti-inflammatory drugs NSAIDS 2 days before (5 days for long-acting NSAIDs), the day of, and 2 days following administration of Pemetrexed.
10. The ability to take folic acid, Vitamin B12, and dexamethasone according to protocol.

Exclusion Criteria:

1. Not pregnant or breastfeeding - the drugs used in this study are Pregnancy Category D (clear evidence of risk in pregnancy). A negative pregnancy test is required within 14 days of registration for pre- or perimenopausal (i.e., last menstrual period within one year of registration) women.
2. Patients with a history of another neoplasm, with the exception of non-metastatic, non-melanoma skin cancers, carcinoma in situ of the cervix, or cancer cured by surgery or small field radiotherapy, within 5 years of registration will be excluded.
3. Patients with uncontrolled cardiovascular disease (a history of hospitalization for acute myocardial infarction, arrhythmia, or congestive heart failure within 3 months prior to registration) will be excluded
4. Registered patients with an active infection or with a fever of ≥ 38.5°C within 24 hours of the first scheduled day of protocol initiation will be excluded until their infection and/or fever resolves.
5. Any other medical condition, including mental illness or substance abuse, deemed by the Investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results.
6. Inability to interrupt use of non-steroidal anti-inflammatory drugs (NSAIDS)
7. Peripheral neuropathy >/= Grade 2 (Common Terminology Criteria for Adverse Events CTCAE)
8. Systemic chemotherapy within 3 weeks of registration
9. Prior Allergies: History of allergic reactions attributed to compounds of similar chemical or biologic composition to cisplatin and pemetrexed
10. Presence of third space fluid which cannot be controlled by drainage.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-09; Primary Completion 2019-09-05 (Actual); Study Completion 2019-09-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with Dose-Limiting Toxicity (DLT) | from the first day of treatment until 4 weeks after the treatment
  Dose limiting toxicity (DLT) is defined as: 1) Grade 4 treatment-related hematologic toxicity that lasts more than for 5 days or grade 3 thrombocytopenia with grade 3 or 4 bleeding, 2) Febrile neutropenia, 3) Grade 3 or greater treatment related non-hematologic toxicity with the following exceptions:Grade 3 diarrhea is a dose limiting toxicity DLT only if the patient was compliant with an anti-diarrheal program consistent with best clinical practice; Grade 3 or 4 nausea and vomiting is a dose limiting toxicity DLT only if the patient was compliant with an antiemetic program consistent with best clinical practice; Alopecia

CONTACTS AND LOCATIONS:
Overall Officials: Shawn Groth, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor St Lukes, Houston, Texas, United States